CLINICAL TRIAL: NCT03243812
Title: Muscle Function and Its Biological and Physiological Determinants in Sickle Cell Disease
Acronym: DREPAMUSCLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL17_0313
Record Dates: First submitted 2017-07-27; First posted 2017-08-09 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Muscle function; Hemorheological disorders
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SS genotype group (Active Comparator): Sickle cell patients with SS genotype. Each subject will undergo the following :
  1. Blood sample
  2. Maximum Voluntary Contraction (MVC) test force before and after a localized muscle endurance test
  3. Localized muscle endurance test: 4 series of 20 submaximal dynamic contractions at 50% of the MVC interspaced with 1 min recovery.
  4. Self-paced six-minute walk test will be conducted according to the guidelines of the American Thoracic Society
  Interventions: Biological: Blood sampling; Other: Maximum Voluntary Contraction (MVC) test force; Other: Localized muscle endurance test; Other: Self-paced six-minute walk test
- SC genotype group (Active Comparator): Sickle cell patients with SC genotype. Each subject will undergo the following :
  1. Blood sample
  2. Maximum Voluntary Contraction (MVC) test force before and after a localized muscle endurance test
  3. Localized muscle endurance test: 4 series of 20 submaximal dynamic contractions at 50% of the MVC interspaced with 1 min recovery.
  4. Self-paced six-minute walk test will be conducted according to the guidelines of the American Thoracic Society
  Interventions: Biological: Blood sampling; Other: Maximum Voluntary Contraction (MVC) test force; Other: Localized muscle endurance test; Other: Self-paced six-minute walk test
- control group (Active Comparator): Healthy subjects. Each subject will undergo the following :
  1. Blood sample
  2. Maximum Voluntary Contraction (MVC) test force before and after a localized muscle endurance test
  3. Localized muscle endurance test: 4 series of 20 submaximal dynamic contractions at 50% of the MVC interspaced with 1 min recovery.
  4. Self-paced six-minute walk test will be conducted according to the guidelines of the American Thoracic Society
  Interventions: Biological: Blood sampling; Other: Maximum Voluntary Contraction (MVC) test force; Other: Localized muscle endurance test; Other: Self-paced six-minute walk test

INTERVENTIONS:
Biological: Blood sampling — Blood sampling will be performed to assess hematological and hemorheological parameters
Other: Maximum Voluntary Contraction (MVC) test force — Maximum Voluntary Contraction (MVC) test force will be performed before and after a localized muscle endurance test
Other: Localized muscle endurance test — Subject will perform 4 series of 20 submaximal dynamic contractions at 50% of the MVC interspaced with 1 min recovery.
Other: Self-paced six-minute walk test — Self-paced six-minute walk test will be conducted according to the guidelines of the American Thoracic Society

SUMMARY:
Background : Sickle cell patients have profound remodeling of their muscle microcirculation networks with signs of amyotrophy. However, the consequences of these muscle alterations on the functional status of muscles are unknown. In addition, whether the poor physical fitness of sickle cell patients can be attributed, at least partly, to an hypothetical muscle dysfunction has never been tested.

Purpose : this study will compare the muscle function of legs between sickle cell patients (SS and SC genotypes) and healthy individuals (AA genotype) before, during and after a short localized muscle endurance exercise.

Abstract : Very recently, a study reported large differences between the muscle microcirculation networks of sickle cell patients compared to healthy individuals with decreased capillary density and higher proportion of large capillaries in the former population. In addition, the same study showed signs of amyotrophy in sickle cell patients. However, the muscle function of sickle cell patients has not been investigated and one may suggest that muscle dysfunction could participate in the decrease of physical fitness, in association with the hematological and hemorheological disorders, already reported in this population. The hypothesis is that muscle fatigue during a short localized muscle endurance exercise should be higher in sickle cell patients compared to healthy individuals, due to a greater recruitment of glycolytic fibers and a faster decrease of muscle oxygenation during exercise.

ELIGIBILITY:
Inclusion Criteria:

For Sickle cell patients :

* age ≥ 15 and < 60 years old,
* SS homozygote or SC heterozygote
* in clinical steady state (i.e. without vaso-occlusive crisis or recent blood transfusion)
* identified by systematic neonatal screening programs,
* registered in the French medical social security national program

For Healthy and non sickle cell subjects:

* age ≥ 18 and < 60 years old
* without cardiovascular/respiratory/muscle disease,
* registered in the French medical social security national program.

Exclusion Criteria:

* other hemoglobinopathies,
* stroke or vasculopathy history,
* presence of leg ulcers or osteonecrosis,
* recent infectious episode (less than 1 month),
* chronic transfusion therapy programs,
* recent blood transfusion or phlebotomies (less than 3 months),
* patients not at steady state,
* pregnancy or breast feeding

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 77 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Maximum isometric muscular strength | Day 1
  Isometric muscular strength will be determined by Maximum Voluntary Contraction (MVC) test force on dominant leg.
  Muscular function will be evaluated using Maximum Voluntary Contraction (MVC) test force and the muscle endurance ability, which will be highlighted by the degree of decline of MVC after a short localized muscle effort using the formula: ((post MVC force - pre MVC force) / pre MVC force)x100.
  Muscle weakness will be determined by a loss of maximum isometric strength ≥ 20 % compared with control group.

SECONDARY OUTCOMES:
Surface Electromyography (EMG) Activity | Day 1
  Surface EMG signals will be recorded by non-invasive electrodes on the dominant leg.
Muscle oxygenation measurement | Day 1
  oxyhemoglobin (HbO2) and deoxyhemoglobin (HHb) levels will be measured using Near-Infrared spectroscopy on the dominant leg.
Measurement of six-minute walk distance (6MWD) | Day 1
  In order to investigate the association between muscle endurance ability and physical fitness in sickle cell patients, patients will realize a six-minute walk test (6MWT).
  6MWD will be measured = the distance that a patient has walked on a flat, hard surface in a period of 6 minutes (6MWT).
Complete Blood Count (CBC) | Day 1
  CBC will be performed in order to evaluate the role of hematological disorders in the muscle fatigue of sickle cell patients.
Hematocrit | Day 1
  Hematocrit will be measured in order to evaluate the role of hematological disorders in the muscle fatigue of sickle cell patients.
Blood viscosity | Day 1
  Blood viscosity will be measured by using viscosimetry, in order to evaluate the role of hemorheological disorders in the muscle fatigue of sickle cell patients.
Red blood cell (RBC) deformability | Day 1
  RBC deformability will be assessed by using ektacytometry, in order to evaluate the role of hemorheological disorders in the muscle fatigue of sickle cell patients.
Aggregation properties | Day 1
  Aggregation properties will be assessed by using syllectometry, in order to evaluate the role of hemorheological disorders in the muscle fatigue of sickle cell patients.
Hemoglobin oxygenation level | Day 1
  Hemoglobin oxygenation level will be measured in order to evaluate the role of hemorheological disorders in the muscle fatigue of sickle cell patients.
Number of vaso-occlusive crises and acute chest syndrome within a 5 years retrospective period. | Day 1
  Number of vaso-occlusive crises and acute chest syndrome reflects of clinical severity of the sickle cell disease.
  Clinical severity will be retrospectively (5 years) collected in clinical record of sickle cell patients.
  These clinical data will be used to study the relationships between the degree of muscle dysfunction and the degree of clinical severity in sickle cell patients.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna CANNAS, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Edouard Herriot, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gouraud E, Connes P, Gauthier-Vasserot A, Faes C, Merazga S, Poutrel S, Renoux C, Boisson C, Joly P, Bertrand Y, Hot A, Cannas G, Hautier C. Is Skeletal Muscle Dysfunction a Limiting Factor of Exercise Functional Capacity in Patients with Sickle Cell Disease? J Clin Med. 2021 May 22;10(11):2250. doi: 10.3390/jcm10112250. PMID 34067352